CLINICAL TRIAL: NCT06415409
Title: Rehydration After Exercise With High-electrolyte Sport Drink
Brief Title: Rehydration Efficiency With Different Sports Drinks
Acronym: REHYDR8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: FP00034719
Record Dates: First submitted 2023-08-23; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Dehydration
MeSH Terms: conditions — Dehydration | interventions — Water; gatorade

STUDY DESIGN:
Intervention Model Description: Randomized Cross over design.
Who Masked: Participant
Masking Description: Unidentified bottles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Water (Placebo Comparator): rehydration with Plain water
  Interventions: Other: Water
- Gatorade (Active Comparator): rehydration with Gatorade drink
  Interventions: Other: Gatorade
- BodyArmor (Active Comparator): Rehydration with Body Armor Drink
  Interventions: Other: BodyArmor
- GoodSport (Experimental): Rehydration with Good Sport drink
  Interventions: Other: GoodSport

INTERVENTIONS:
Other: Water — Plain water
  Arms: Water
Other: Gatorade — Sport Drink Gatorade
  Arms: Gatorade
Other: BodyArmor — Sport Drink BodyArmor
  Arms: BodyArmor
Other: GoodSport — Sport Drink GoodSport
  Arms: GoodSport

SUMMARY:
It is well established that post-exercise rehydration with a carbohydrate-electrolyte solution is better when compared to plain water. However, most of the commercially available drinks today are high in carbohydrates and sodium with low potassium without other active ingredients. The aim of the present study is to examine the impact of a higher electrolyte sports drink compared with traditional sports drinks and water on the time course and extent of rehydration after exercise-induced dehydration

DETAILED DESCRIPTION:
Dehydration:

Based on our previous work, dehydration will be accomplished on the morning of testing via mild exercise and heat exposure to elicit a body weight loss of -2%. The subjects will perform four bouts of 25-min low-intensity exercise and 5 min rest (alternating cycling & walking) or till they reach -2% of body weight dehydration.

Rehydration:

Following a 20 min rest in thermo-comfortable environment a dehydrated baseline blood sample will be taken, and subject will start the rehydration protocol.

The volunteers will consume one of the four drinks below in a cross over balance mode. During the first hour four equal doses will be consumed in15-min intervals at a total volume of 150% of their body weight loss.

Trials/Drinks (block randomization will be used to assign individual participants to each specific trial/drink using their ID number):

* Water
* GoodSport®
* Gatorade®
* BodyArmor®

Measurements:

All measurements will be performed at one of the test rooms at our lab facility that boarders the room where participants can relax and wait out the end of the study day. When certain measurements need to be performed they simply move from one room to the next. Duration of taking blood and urine samples will take not more than 30-90 seconds each, bioelectrical impedance will take a bit more time to ensure the body is in a stable rested state as a result measurement will be taken in 10 minutes, finally perceptual data will take 30-60 seconds to be reported. To allow to perform all measurements study days will take up to 7 hours. Therefore, there will be a separate space available that allows for self-study or watching TV that includes a chair and table to work on and a couch to relax.

Blood samples (8 per trial, maximal 12 minutes):

A total of eight 10 mL blood samples will be collected on the euhydrated baseline, dehydrated baseline and at 30, 60, 90, 120, 180, and 240 min of the rehydration period.

All samples will be analyzed for glucose, osmolality, total plasma protein, hematocrit, hemoglobin (for plasma volume changes), sodium, potassium, and chloride.

Urine samples (6 per trial, maximal 9 minutes):

Urine samples will be collected using ~900 mL cups at euhydrated baseline, dehydrated baseline and cumulative totals will be collected at 60, 120, 180, and 240 min of the rehydration period. All samples will be analyzed for urine osmolality, specific gravity, volume, sodium, and potassium.

Perceptual Data (6 per trial, maximal 9 minutes):

Thirst, stomach fullness, and taste, assessed via a visual analog scale

ELIGIBILITY:
Inclusion Criteria:

* Training > 2x per week
* Age 18-55 y
* stable weight for the last 2 months (<5 lbs. fluctuation)

Exclusion Criteria:

* night shifting work
* thyroid medication
* bariatric surgery
* cardiovascular disease
* renal disease
* hepatic disease
* Participating in another study at the same time
* Bodyweight <110 lbs.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Net Fluid Balance | 3 hours of rehydration
  Net fluid balance based on body weight changes during the 4 h of the rehydration period
Net Fluid Balance | 4 hours of rehydration
  Net fluid balance based on body weight changes during the 4 h of the rehydration period
Urine volume | 3 hours of rehydration
  cumulative Urine output during the rehydration period
Urine osmotic excretion | 3 hours of rehydration
  Urine osmotic excretion during rehydration
Urine osmotic excretion | 4 hours of rehydration
  Urine osmotic excretion during rehydration

SECONDARY OUTCOMES:
Stomach fullness | 3 hours of rehydration
  Assessed via a Visual Analog scale during rehydration
Stomach fullness | 4 hours of rehydration
  Assessed via a Visual Analog scale during rehydration. Scale is from 0-125mm with higher number indicating greater perception
Thirst | 3 hours of rehydration
  Assessed via a Visual Analog scale during rehydration. Scale is from 0-125mm with higher number indicating greater perception
Thirst | 4 hours of rehydration
  Assessed via a Visual Analog scale during rehydration. Scale is from 0-125mm with higher number indicating greater perception

CONTACTS AND LOCATIONS:
Locations (1):
- Interdisciplinary Science and Technology Building 8, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No